CLINICAL TRIAL: NCT04077619
Title: Shifting Away From Pain: Neurocognitive Approach to Explain and Predict the Response to the Modern Neuroscience Approach for Treating Patients With Whiplash Associated Disorders
Brief Title: Shifting Away From Pain: a Neurocognitive Approach in Treatment of Whiplash
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B143201630602; G001419N (Other Grant/Funding Number: Research Foundation Flanders)
Record Dates: First submitted 2019-08-22; First posted 2019-09-04 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Whiplash Injuries
MeSH Terms: conditions — Whiplash Injuries

STUDY DESIGN:
Intervention Model Description: The other trial (NCT03239938) will randomize patients with chronic WAD to the experimental (modern neuroscience approach) or the control treatment (usual care physiotherapy). The WAD patient sample for the present MRI study will be a subsample recruited from this larger RCT. After inclusion in the large RCT, participants will be asked about the possibility of participating in the additional MRI study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modern pain neuroscience approach (Experimental): Behavioral: Modern pain neuroscience approach
  Interventions: Behavioral: Modern pain neuroscience approach
- Usual care evidence-based physiotherapy (Active Comparator): Behavioral: Usual care evidence-based physiotherapy
  Interventions: Behavioral: Usual care physiotherapy

INTERVENTIONS:
Behavioral: Modern pain neuroscience approach — Modern pain neuroscience approach. The modern pain neuroscience approach includes 3 sessions (1 group and 2 individual sessions) of therapeutic pain neuroscience education followed by 15 individual sessions of dynamic and functional cognition-targeted exercise therapy and stress management techniques. In addition, participants will be instructed to perform a daily set of home exercises. The exercises will be performed in a time-contingent way. The 18 sessions will be spread over a period of 16 weeks.
  Arms: Modern pain neuroscience approach
Behavioral: Usual care physiotherapy — Usual care evidence-based physiotherapy The usual care evidence-based physiotherapy includes 3 sessions (1 group and 2 individual sessions) of neck school followed by 15 individual sessions of graded and active exercise therapy focusing on strength, flexibility, endurance, and ergonomic principles. In addition, participants will be instructed to perform a daily set of home exercises. The exercises will be performed in a symptom-contingent way. The 18 sessions will be spread over a period of 16 weeks.
  Arms: Usual care evidence-based physiotherapy

SUMMARY:
The broad aim of this study is to investigate the effect of a modern neuroscience approach, which combines education on pain neuroscience with cognition-targeted exercise therapy and stress management, on brain structure and networks in patients with chronic whiplash-associated disorders (CWAD) in comparison to a control physiotherapy treatment.

DETAILED DESCRIPTION:
This project runs in parallel to a larger randomized-controlled trial (RCT) in which the 'modern neuroscience approach to WAD' is compared to usual care evidence-based physiotherapy (clinical trial registration number: NCT03239938). For the current study, additional magnetic resonance imaging (MRI) measures will be taken in a subsample of patients, who will be recruited from this larger RCT. In addition, a pain-free age- and sex-matched control group will be recruited for comparison.

The current study consists of 2 MRI measurements that will take place at the University Hospital of Ghent (UZ Gent): baseline (pre-treatment) and follow-up (post-treatment; approximately 16 weeks after baseline). After pre-treatment assessment, the patients will be randomly allocated to the modern neuroscience approach or usual care physiotherapy, as part of the RCT.

ELIGIBILITY:
CWAD group:

Inclusion Criteria:

* Experienced a whiplash trauma which is at least 3 months old and causes pain since at least 3 months, with pain experience with a mean pain frequency of 3 or more days per week, and with self-reported moderate to severe pain-related disability, established by a score of 15 or more of a maximum of 50 on the Neck Disability Index
* Patients classified as WAD II or WAD III on the modified Quebec Task Force Scale
* Native Dutch speaker
* Not starting new treatments or medication and continuing their usual care 6 weeks prior to and during study participation (to obtain a steady state)
* Refraining from consuming caffeine, alcohol and nicotine in the hour before the MRI scans (in both measurement times: before the start of the rehabilitation and after the end of the rehabilitation).

Exclusion Criteria:

* Neuropathic pain
* Being pregnant or having given birth in the preceding year
* Chronic fatigue syndrome
* Fibromyalgia
* Cardiovascular disorders
* Epilepsy
* Endocrinological disorders
* Rheumatic disorders
* Psychiatric disorders
* History of neck surgery
* Loss of consciousness during/after the whiplash trauma
* MRI incompatible health condition (e.g., pacemaker, metal prosthetic devices)
* Psychiatric condition and ongoing medication that would alter emotional or sensory processing
* Claustrophobia.

Healthy volunteers: (matched for age and gender). Additional exclusion criteria include for healthy volunteers

* a history of a chronic pain syndrome
* a pain condition in the last six months for which treatment was sought

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
blood oxygenation level dependent (BOLD) signal (functional MRI) during picture imagination task and during resting state | Baseline (pre-treatment) assessment and follow-up assessment after 16 weeks of therapy (end of treatment).
  change between baseline assessment and the follow-up assessment after 16 weeks (after end of treatment) will be examined
structural MRI measures (i.e., grey and white matter) | Baseline (pre-treatment) assessment and follow-up assessment after 16 weeks of therapy (end of treatment).
  change between baseline assessment and the follow-up assessment after 16 weeks (after end of treatment) will be examined

CONTACTS AND LOCATIONS:
Overall Officials: Mira Meeus, PhD, Principal Investigator — University Ghent; Iris Coppieters, PhD, Study Director — University Ghent
Locations (1):
- Department of rehabilitation sciences (Ghent University), Ghent, Belgium